CLINICAL TRIAL: NCT01929317
Title: A Study ROP116991, Clinical Evaluation of 18 to 24mg/Day Ropinirole CR for Parkinson's Disease.
Brief Title: A Study to Evaluate the Efficacy of 18 to 24mg/Day Ropinirole Controlled Release (CR) Tablets in Early and Advanced Parkinson's Disease (PD) Patients.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116991
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
Keywords: Ropinirole; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropinirole CR high-dose group (Experimental): The subjects will receive Ropinirole CR 16mg/day for 4 weeks in screening phase. After randomization the subject will enter dose increase effect verification phase, where Ropinirole CR dose will titrated (2 mg /day/week) from 18 mg/day up to a maximum 24mg/day at intervals of 1 week or longer for 8 weeks, till subject reaches a dose level above which further symptomatic improvement cannot be expected; the subject will be maintained on that dose for 4 weeks. This will be followed by a down titration phase of one week and long term phase of 39 weeks in which the subjects will receive incremental doses (2 mg /day/week) of Ropinirole CR from 18 mg/day till to a maximum of 24 mg/day till subject reaches a dose level above which further symptomatic improvement cannot be expected; the subject will be maintained on that dose. Subjects completing the long term phase will undergo a down titration phase of 1 to 2 weeks.
  Interventions: Drug: Ropinirole CR 2mg tablet; Drug: Ropinirole CR 8mg tablet
- Ropinirole CR maintenance group (Experimental): The subjects will receive Ropinirole CR 16mg/day for 4 weeks in screening phase. After randomization the subject will enter dose increase effect verification phase and Ropinirole CR dose will maintained at 16mg/day and placebo will be increased at intervals of 1 week for 8 weeks till subject reaches a dose level above which further symptomatic improvement cannot be expected; the subject will be maintained on that dose for 4 weeks. This will be followed by a down titration phase of one week and long term phase of 39 weeks in which the subjects will receive incremental doses (2 mg/day/week) of Ropinirole CR from 18 mg/day till to a maximum of 24 mg/day till subject reaches a dose level above which further symptomatic improvement cannot be expected; the subject will be maintained on that dose. Subjects completing the long term phase will undergo a down titration phase of 1 to 2 weeks.
  Interventions: Drug: Ropinirole CR 2mg tablet; Drug: Ropinirole CR 8mg tablet; Drug: Ropinirole CR matching Placebo tablet

INTERVENTIONS:
Drug: Ropinirole CR 2mg tablet — Ropinirole CR 2mg tablets will be supplied as white oval film-coated tablets.
Drug: Ropinirole CR 8mg tablet — Ropinirole CR 8mg tablets will be supplied as white oval film-coated tablets.
Drug: Ropinirole CR matching Placebo tablet — Ropinirole CR matching Placebo tablet tablets (containing no active ingredients) indistinguishable in appearance from Ropinirole CR 2 mg tablets.
  Arms: Ropinirole CR maintenance group

SUMMARY:
This study is a Phase III, multicentre, randomized, initial double-blind study with subsequent open label phases. The study will havea screening phase (4 weeks), a dose increase effect verification phase (12 weeks), a down titration 1 phase (1 week), a long-term phase (39 weeks), down titration 2 phase (1 to 2 weeks) and a follow up phase. Subjects will be assigned to Ropinirole CR high-dose group or Ropinirole CR maintenance group at a ratio of 3:1. This study is being conducted to evaluate the efficacy (effect of increasing Ropinirole dose from 16 mg/day to 18-24 mg/day) of the Ropinirole CR tablets in early and advanced PD patients who have not achieved an optimal therapeutic response with marketed Ropinirole Immediate release (IR) (15 mg/day) or marketed Ropinirole CR (16 mg/day) formulations.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria at the start of the screening

* Patients who are diagnosed as Parkinson's Disease with severity of the modified Hoehn & Yahr criteria Stages I-IV.
* 1) Monotherapy subject: Subjects who have never received L-dopa, or subjects who have had prior exposure to L-dopa (up to 450 milligram (mg)/day) for up to 3 months in total and L-dopa treatment has been discontinued, for a minimum of 4 weeks prior to the screening phase. 2) L-dopa adjunct subject: Subjects receiving L-dopa (up to 450 mg/day) for at least 4 weeks prior to the screening phase.
* Patients receiving 15mg/day Ropinirole IR or 16mg/day Ropinirole CR for 4 weeks prior to the screening phase, UPDRS Part III total (on) scores is 10 points or more at screening visit and can expect clinical efficacy by increasing Ropinirole CR.
* Age: 20years or older (at the time of informed written consent)
* Informed consent: Patients who are able to give informed written consent in person. (i.e. patients who are capable of giving informed written consent on their own)
* Sex: Either sex. Women of child-bearing potential will be eligible for inclusion in this study. However they have to have a negative pregnancy test at the screening visit and will have to agree to further pregnancy testing at the time points determined in study assessments and procedures and practice one of the methods of contraception mentioned in the protocol from the screening visit until the end of the follow-up examination - Outpatient status
* corrected QT (QTc) <450 millisecond (msec) or <480msec for subjects with Bundle Branch Block. The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* Liver function tests: Patients with aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2x upper limit of normal (ULN); and Alkaline Phosphatase and bilirubin =< 1.5xULN (isolated bilirubin > 1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) at the screening visit.

Randomization Criteria

* Patients whose UPDRS Part III total (on) scores is 10 points or more at week 0
* Patients who did not achieve an optimal therapeutic response by treatment with 16mg/day Ropinirole CR and required higher dose of Ropinirole CR
* Patients who are 80% or more compliant taking study drug

Exclusion Criteria

* Late stage advanced patients demonstrating incapacitating peak dose or biphasic dyskinsia on their stable dose of L-dopa.
* Patients who have used any other dopamine agonist (except for Ropinirole IR and CR) within 4 weeks prior to the screening phase.
* Patients who have been treated with the following drugs at 4 weeks or earlier before the start of the screening phase, and whose treatment regimen of the drug has been changed. Anticholinergic agents: trihexyphenidyl hydrochloride, piroheptine hydrochloride, mazaticol hydrochloride, metixene hydrochloride, biperiden hydrochloride, profenamine, amantadine hydrochloride,droxidopa, citicoline, selegiline hydrochloride, entacapone, zonisamide, Estrogens, CYP1A2 inhibitors.
* Patients who have been changing in smoking habit (started or stopped smoking) within the screening phase.
* Patients who have been treated with any other investigational drug within 12 weeks prior to the screening phase.
* Patients who present serious physical signs and symptoms other than those of the PD (e.g. cardiac/hepatic/renal disorder and haematopoietic disorder).
* Patients with symptomatic postural hypotension. (e.g. dizziness and syncope).
* Patients with a current or history of drug abuse or alcoholism.
* Patients with severe dementia such as score 3 or 4 of the UPDRS item 1 (Mentation, behaviour, and mood).
* Patients with current or history of major psychosis (e.g. schizophrenia or psychotic depression) such as score 3 or 4 of the UPDRS item 2 (thought disorder) or item 3(depression).
* Patients who have received surgical treatment for PD in the past (e.g. pallidectomy, deep brain stimulation).
* Female patients who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study or within 30 days after the last dose of the study drug.
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulapathy, hypoalbuminaemia, oesophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Chronic hepatitis B administered immunosuppressive agents due to risk of hapatitis B reactivation.
* Patients with a history of drug allergy to Ropinirole hydrochloride.
* Except for patients with a history of basal cell carcinoma, patients with a current or history of cancer or malignant tumor within 5 years prior to the screening phase.
* Others whom the investigator (subinvestigator) considers ineligible for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2014-09-16 (Actual); Study Completion 2015-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Japan (12):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Akita
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hattori N, Hasegawa K, Sato K, Mitsuyama E, Numachi Y. Clinical evaluation of ropinirole controlled-release formulation at 18-24 mg/day in Japanese patients with Parkinson's disease. Parkinsonism Relat Disord. 2017 Jul;40:33-39. doi: 10.1016/j.parkreldis.2017.04.005. Epub 2017 Apr 13. PMID 28442303
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 116991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116991 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 81 participants (par.) were randomized, of which 71 participants completed the Dose Increase Effect Verification (DIEV) Phase and 62 participants entered the Long-term Phase and 39 participants completing the Long-term Phase.
Pre-assignment Details: This study was comprised of a Screening Phase (4 weeks), DIEV Phase (12 weeks), Down Titration 1 Phase (1 week), Long-term Phase (39 weeks), Down Titration 2 Phase (1 to 2 weeks) and the Follow-up Phase. The first 60 par. who completed the DIEV phase entered into the Long-term phase after a completion of the Down Titration 1 phase.
Groups:
- Ropinirole CR - High Dose Group: Participants received ropinirole controlled released (CR) 16 milligrams (mg) administered orally once daily (OD) for 4 weeks in the Screening Phase. After randomization, participants entered the Dose Increase Effect Verification Phase, where ropinirole CR dose was titrated (2 mg/day/week) from 18 mg/day up to a maximum 24 mg/day at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. After the completion of the Dose Increase Effect Verification Phase, participants entered the Down Titration Phase for 1 week and selected participants entered the Long-term Phase for 39 weeks.
- Ropinirole CR - Maintenance Dose Group: Participants received ropinirole CR 16 mg per day administered orally OD for 4 weeks in the Screening phase. After randomization, participants entered the Dose Increase Effect Verification Phase, where ropinirole CR dose was maintained at 16 mg/day and the placebo was titrated to maintain blinding at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. After the completion of the Dose Increase Effect Verification Phase, participants entered the Down Titration Phase for 1 week and selected participants entered the Long-term Phase for 39 weeks.
Period: Dose Increase Effect Verification Phase
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Started | 61 | 20
Completed | 52 | 19
Not Completed | 9 | 1
Not completed — Adverse Event | 5 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Period: Long-term Phase
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Started | 44 | 18
Completed | 25 | 14
Not Completed | 19 | 4
Not completed — Adverse Event | 5 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0
Not completed — Study Closed/Terminated | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Ropinirole CR - High Dose Group: Participants received ropinirole CR 16 mg administered orally OD for 4 weeks in the Screening Phase. After randomization the participant entered Dose Increase Effect Verification Phase, where Ropinirole CR dose was titrated (2 mg/day/week) from 18 mg/day up to a maximum 24mg/day at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. This was followed by a down titration phase for one week and Long-term Phase for 39 weeks in which the participants received incremental doses (2 mg/day/week) of ropinirole CR from 18 mg/day to a maximum of 24 mg/day until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose. Participants completed the Long-term Phase underwent a down titration phase 2 for 1 to 2 weeks.
- Ropinirole CR - Maintenance Dose Group: Participants received ropinirole CR 16 mg administered orally OD for 4 weeks in the Screening Phase. After randomization participants entered Dose Increase Effect Verification Phase, where Ropinirole CR dose was maintained at 16 mg/day and the placebo was titrated to maintain blinding at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. This was followed by a down titration phase for one week and Long-term Phase for 39 weeks in which the participants received incremental doses (2 mg/day/week) of ropinirole CR from 18 mg/day to a maximum of 24 mg/day until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose. Participants completed the Long-term Phase underwent a down titration phase 2 for 1 to 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group | Total
Number analyzed (Participants) | 61 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (8.95) | 63.3 (12.42) | 65.0 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 11 | 50
  Male | 22 | 9 | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese/East Asian Heritage (EAH)/South EAH | 61 | 20 | 81

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Week 0) in UPDRS Part III Total Score at Week 12 in the CR High-dose Group
Description: The Japanese Unified Parkinson's Disease Rating Scale (UPDRS) assesses the status of Parkinson's Disease (PD) participants objectively. Part III assessed motor examination on 27 items. Participants received a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. Baseline is defined as the value evaluated at Week 0. Mean change from Baseline was calculated as the total score at Week 12 minus the total score at Baseline. The analyses for the Dose Increase Effect Verification Phase was performed using the last observation carried forward (LOCF) data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit. The imputation was conducted using the data within only the Dose Increase Effect Verification Phase; therefore, the value observed in the Dose Increase Effect Verification Phase was not used to impute a missing data in the Long-term Phase.
Time Frame: Baseline and Week 12
Population: Full Analysis Set 1 (FAS1) Population: all participants excluding those participants who received no dose of study medication and participants without UPDRS part III total score data after supply of the investigational product.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group
Number analyzed (Participants) | 61
Scores on a scale | -4.8 (5.95)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; Mean change from Baseline = -4.8, 95% CI 2-sided [-6.3 to -3.2]

2. Secondary Outcome: Mean Change From Baseline (Week 0) in UPDRS Part III Total Score at the Indicated Visits
Description: as for outcome 1
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Scores on a scale
  Week 2 | -2.9 (4.41) | -2.7 (4.27)
  Week 4 | -3.8 (5.23) | -4.4 (3.50)
  Week 6 | -4.6 (5.28) | -5.0 (5.09)
  Week 8 | -5.2 (5.46) | -4.5 (4.94)
  Week 12 | -4.8 (5.95) | -5.7 (5.18)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.4 to 2.0] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part III total score for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.9 to 3.1] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part III total score for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.3 to 3.0] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part III total score for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.4 to 2.0] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part III total score for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.0 to 3.9] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part III total score for Week 12

3. Secondary Outcome: Number of Participants Achieving a 30% and 20% Reduction From Baseline in the UPDRS Total Part 3 Score at the Indicated Visits in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assesses the status of Parkinson's Disease (PD) participants objectively. Part III assessed motor examination on 27 items. Participants received a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. Number of participants achieving a 30% or greater and 20% or greater reduction from Baseline in UPDRS total part III score at Weeks 2, 4, 6, 8, and 12 are presented using LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit. The imputation was conducted using the data within only the Dose Increase Effect Verification Phase; therefore, the value observed in the Dose Increase Effect Verification Phase was not used to impute a missing data in the Long-term Phase.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Participants
  Week 2, 30% or greater reduction from Baseline | 10 | 4
  Week 4, 30% or greater reduction from Baseline | 17 | 5
  Week 6, 30% or greater reduction from Baseline | 21 | 6
  Week 8, 30% or greater reduction from Baseline | 30 | 7
  Week 12, 30% or greater reduction from Baseline | 27 | 7
  Week 2, 20% or greater reduction from Baseline | 16 | 5
  Week 4, 20% or greater reduction from Baseline | 26 | 11
  Week 6, 20% or greater reduction from Baseline | 30 | 10
  Week 8, 20% or greater reduction from Baseline | 35 | 11
  Week 12, 20% or greater reduction from Baseline | 31 | 13

4. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part 1 Total Score at the Indicated Visits in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part I evaluated mentation, behavior, and mood on 4 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 16. A higher score indicates more severe PD symptoms. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 0. The analyses for the Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at the planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Scores on a scale
  Week 2 | -0.0 (0.50) | -0.1 (0.31)
  Week 4 | -0.1 (0.57) | -0.2 (0.49)
  Week 6 | -0.1 (0.69) | -0.1 (0.45)
  Week 8 | -0.1 (0.68) | -0.1 (0.45)
  Week 12 | 0.1 (0.89) | -0.1 (0.45)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.3] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 1 total score for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.2 to 0.4] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 1 total score for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.3] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 1 total score for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.3] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 1 total score for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 1 total score for Week 12

5. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part 2 Total Score at the Indicated Visits by the on/Off Status in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part 2 evaluated activities of daily living on 13 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 52. A higher score indicates more severe PD symptoms. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 0. The analyses for the Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "On" state is defined as the state at which PD symptoms are well controlled by the drug. The score of UPDRS part 2 in off status is rated as '0' (Normal/None), if L-dopa adjunct participants do not have diurnal fluctuations.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the FAS1 population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Scores on a scale
  Week 2, On status, n=61, 20 | -1.0 (2.00) | -0.2 (0.99)
  Week 4, On status, n=61, 20 | -1.4 (2.60) | -0.3 (1.63)
  Week 6, On status, n=61, 20 | -1.6 (3.03) | -0.5 (2.04)
  Week 8, On status, n=61, 20 | -1.4 (3.23) | -0.2 (2.23)
  Week 12, On status, n=61, 20 | -1.1 (3.61) | -0.2 (2.64)
  Week 2, Off status, n=53, 18 | -1.0 (2.13) | -0.3 (1.97)
  Week 4, Off status, n=53, 18 | -1.3 (3.23) | -0.4 (2.89)
  Week 6, Off status, n=53, 18 | -1.7 (3.90) | -0.8 (2.26)
  Week 8, Off status, n=53, 18 | -1.4 (3.92) | -1.3 (2.27)
  Week 12, Off status, n=53, 18 | -1.4 (4.25) | -1.3 (2.52)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.8 to 0.1] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 2, On status
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.4 to 0.1] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 4, On status
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.6 to 0.3] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 6, On status
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.8 to 0.3] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 8, On status
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.7 to 0.7] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 12, On status
Statistical Analysis 6: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.8 to 0.5] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 2, Off status
Statistical Analysis 7: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.6 to 0.8] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 4, Off status
Statistical Analysis 8: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.8 to 1.0] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 6, Off status
Statistical Analysis 9: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.1 to 1.8] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 8, Off status
Statistical Analysis 10: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.2 to 2.1] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 2 total score for Week 12, Off status

6. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part 4 Total Score at the Indicated Visits in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part 4 evaluated complications on 11 items, response for 4 items were scored numerically from 0-4 and response for other 7 items were Yes/No questions and responses are numerically scored as 0 for "No" and 1 for "Yes". The total score for the 11 items ranged from 0 to 23. A higher score indicates more severe PD symptoms. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 0. The analyses for the Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Scores on a scale
  Week 2 | -0.3 (1.10) | -0.2 (1.01)
  Week 4 | -0.2 (1.24) | -0.2 (1.39)
  Week 6 | -0.2 (1.43) | -0.3 (1.49)
  Week 8 | 0.0 (1.32) | 0.1 (1.28)
  Week 12 | -0.1 (1.38) | 0.1 (1.29)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.4] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 4 total score for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.6] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 4 total score for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.7 to 0.8] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 4 total score for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 4 total score for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.5] — Estimated value and CI are presented for the change from Baseline in Japanese UPDRS Part 4 total score for Week 12

7. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 1 Total Score at the Indicated Visits in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part I evaluated mentation, behavior, and mood on 4 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 16. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value evaluated at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 21 | 8
Percent change
  Week 2 | -6.2 (40.06) | -16.7 (35.63)
  Week 4 | -14.5 (63.87) | -41.7 (49.60)
  Week 6 | -15.2 (83.82) | -29.2 (45.21)
  Week 8 | -16.4 (82.27) | -29.2 (45.21)
  Week 12 | -7.4 (85.84) | -29.2 (45.21)

8. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 2 Total Score at the Indicated Visits by the on/Off Status in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part 2 evaluates activities of daily living on 13 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 52. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit. "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "On" state is defined as the state at which PD symptoms are well controlled by the drug. The score of UPDRS part 2 in off status is rated as '0' (Normal/None), if L-dopa adjunct participants do not have diurnal fluctuations.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Percent change
  Week 2, On status, n=55, 16 | -22.3 (35.46) | -4.6 (20.29)
  Week 4, On status, n=55, 16 | -21.9 (43.38) | -13.0 (39.07)
  Week 6, On status, n=55, 16 | -21.4 (48.64) | -12.9 (53.71)
  Week 8, On status, n=55, 16 | -14.3 (75.53) | -9.0 (59.34)
  Week 12, On status, n=55, 16 | -4.7 (102.75) | -9.3 (63.12)
  Week 2, Off status, n=48, 15 | -11.7 (26.38) | -4.2 (13.45)
  Week 4, Off status, n=48, 15 | -15.0 (36.35) | -4.4 (18.18)
  Week 6, Off status, n=48, 15 | -17.0 (42.27) | -9.7 (17.69)
  Week 8, Off status, n=48, 15 | -14.7 (40.53) | -10.9 (16.68)
  Week 12, Off status, n=48, 15 | -15.2 (44.90) | -10.1 (14.02)

9. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 3 Total Score at the Indicated Visits in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part 3 evaluated motor examination on 27 items, response for each items were scored numerically from 0-4. The total score for the 27 items ranged from 0 to 108. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value evaluated at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 61 | 20
Percent change
  Week 2 | -12.0 (18.69) | -11.8 (22.78)
  Week 4 | -17.4 (23.29) | -21.9 (18.81)
  Week 6 | -21.6 (23.96) | -22.9 (23.74)
  Week 8 | -25.5 (26.97) | -22.9 (25.02)
  Week 12 | -23.1 (29.88) | -27.6 (28.37)

10. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 4 Total Score at the Indicated Visits in the Dose Increase Effect Verification Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part 4 evaluated complications on 11 items, response for 4 items were scored numerically from 0-4 and response for other 7 items were Yes/No questions and responses are numerically scored as 0 for "No" and 1 for "Yes". The total score for the 11 items ranged from 0 to 23. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value evaluated at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 54 | 19
Percent change
  Week 2 | -7.9 (36.71) | -1.9 (31.59)
  Week 4 | -4.1 (41.73) | -6.5 (35.97)
  Week 6 | -7.2 (47.39) | -4.9 (36.92)
  Week 8 | 1.4 (46.48) | 3.5 (35.18)
  Week 12 | -6.6 (46.04) | 9.5 (30.44)

11. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part 1 Total Score at the Indicated Visits in the Long-term Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part I evaluated mentation, behavior, and mood on 4 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 16. A higher score indicates more severe PD symptoms.Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data. Full Analysis Set 2 (FAS2) Population comprised of all participants in the FAS1 and shifted to Long-term Phase, excluding those participants who received no dose of study medication and participants without UPDRS part III total score data after supply of the investigational product.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: FAS2 Population. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the FAS2 population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ropinirole CR - High Dose Group: Long Term Phase; Ropinirole CR - Maintenance Group: Long Term Phase: Participants received ropinirole CR 16 mg administered orally OD for 4 weeks in the Screening Phase. After randomization the participant entered Dose Increase Effect Verification Phase, where Ropinirole CR dose was titrated (2 mg/day/week) from 18 mg/day up to a maximum 24mg/day at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. This was followed by a down titration phase for one week and Long-term Phase for 39 weeks in which the participants received incremental doses (2 mg/day/week) of ropinirole CR from 18 mg/day to a maximum of 24 mg/day until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose. Participants completed the Long-term Phase underwent a down titration phase 2 for 1 to 2 weeks.
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Scores on a scale
  Week 17; n=42,17 | 0.1 (0.45) | 0.1 (0.56)
  Week 21; n=40, 16 | 0.2 (0.88) | -0.2 (0.66)
  Week 25; n=40, 17 | 0.2 (0.86) | -0.1 (0.83)
  Week 37; n=33, 17 | 0.2 (1.02) | 0.1 (0.90)
  Week 49; n=26, 14 | 0.2 (0.51) | 0.1 (0.73)
  Week 52; n=25, 14 | 0.2 (0.58) | 0.2 (0.97)

12. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part 2 Total Score at the Indicated Visits by the on/Off Status in the Long Term Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part 2 evaluates activities of daily living on 13 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 52. A higher score indicates more severe PD symptoms.Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value at Week 13. If the value at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data."Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "On" state is defined as the state at which PD symptoms are well controlled by the drug. The score of UPDRS part 2 in off status is rated as '0' (Normal/None), if L-dopa adjunct participants do not have diurnal fluctuations.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ropinirole CR - Maintenance Group: Long Term Phase: Participants received ropinirole CR 16 mg administered orally OD for 4 weeks in the Screening Phase. After randomization participants entered Dose Increase Effect Verification Phase, where Ropinirole CR dose was maintained at 16 mg/day and the placebo was titrated to maintain blinding at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. This was followed by a down titration phase for one week and Long-term Phase for 39 weeks in which the participants received incremental doses (2 mg/day/week) of ropinirole CR from 18 mg/day to a maximum of 24 mg/day until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose. Participants completed the Long-term Phase underwent a down titration phase 2 for 1 to 2 weeks.
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Scores on a scale
  Week 17, On status, n=42, 17 | -0.1 (1.52) | 0.1 (0.60)
  Week 21, On status, n=40, 16 | -0.4 (1.60) | 0.0 (0.89)
  Week 25, On status, n=40, 17 | -0.2 (1.91) | -0.1 (0.99)
  Week 37, On status, n=33, 17 | 0.0 (2.32) | 0.2 (1.48)
  Week 49, On status, n=26, 14 | 0.0 (2.41) | 0.6 (1.70)
  Week 52, On status, n=25, 14 | -0.2 (2.67) | 0.1 (1.35)
  Week 17, Off status, n=36, 15 | -0.4 (2.33) | -0.5 (1.46)
  Week 21, Off status, n=34, 14 | -0.4 (2.32) | -0.7 (1.07)
  Week 25, Off status, n=34, 15 | -0.2 (2.27) | -1.5 (3.14)
  Week 37, Off status, n=29, 15 | 0.9 (3.77) | 0.0 (5.01)
  Week 49, Off status, n=24, 12 | 0.4 (3.11) | 0.8 (4.84)
  Week 52, Off status, n=23, 12 | 0.4 (2.52) | 0.8 (4.32)

13. Secondary Outcome: Mean Change From Baseline in UPDRS Part 3 Total Score at the Indicated Visits for Long Term Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part 3 evaluates motor examination on 27 items, response for each items were scored numerically from 0-4. The total score for the 27 items ranged from 0 to 108. A higher score indicates more severe PD symptoms. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49, 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Scores on a scale
  Week 17; n=41, 16 | -1.2 (3.46) | -0.7 (5.03)
  Week 21, n=39, 16 | -2.5 (5.53) | -1.9 (4.92)
  Week 25, n=40, 17 | -2.1 (5.09) | -0.6 (4.31)
  Week 37; n=33, 17 | -1.9 (6.46) | 1.4 (7.65)
  Week 49; n=26, 14 | -2.2 (8.66) | 0.6 (7.38)
  Week 52; n=25, 14 | -1.9 (6.92) | -0.6 (5.49)

14. Secondary Outcome: Change From Baseline in the Japanese UPDRS Part 4 Total Score at the Indicated Visits in the Long Term Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part 4 evaluated complications on 11 items, response for 4 items were scored numerically from 0-4 and response for other 7 items were Yes/No questions and responses are numerically scored as 0 for "No" and 1 for "Yes". The total score for the 11 items ranged from 0 to 23. A higher score indicates more severe PD symptoms.Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Scores on a scale
  Week 17, n=42, 17 | 0.1 (0.97) | -0.1 (1.03)
  Week 21, n=40, 16 | 0.3 (1.01) | -0.1 (0.89)
  Week 25, n=40, 17 | 0.4 (0.83) | 0.2 (2.24)
  Week 37; n=33;17 | 0.5 (1.15) | 1.1 (2.80)
  Week 49; n=26,14 | 0.9 (1.28) | 1.2 (2.72)
  Week 52; n=25, 14 | 0.6 (1.04) | 0.8 (2.36)

15. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 1 Total Score at the Indicated Visits in the Long Term Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part I evaluated mentation, behavior, and mood on 4 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 16. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Percent change
  Week 17, n=15, 7 | 13.3 (36.43) | -9.5 (71.27)
  Week 21, n=14, 7 | -7.1 (28.47) | -31.0 (53.08)
  Week 25, n=14, 7 | 3.6 (48.89) | -26.2 (60.75)
  Week 37; n=9, 7 | 0.0 (43.30) | -11.9 (77.41)
  Week 49; n=6, 5 | 20.8 (40.05) | 15.0 (85.88)
  Week 52; n=6, 5 | 12.5 (44.02) | 5.0 (75.83)

16. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 2 Total Score at the Indicated Visits by the on/Off Status in the Long-term Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part 2 evaluates activities of daily living on 13 items, response for each item were scored numerically from 0-4. The total score for the 4 items ranged from 0 to 52. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value at Week 13. If the value at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data."Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. "On" state is defined as the state at which PD symptoms are well controlled by the drug. The score of UPDRS part 2 in off status is rated as '0' (Normal/None), if L-dopa adjunct participants do not have diurnal fluctuations.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Percent change
  Week 17, On status, n=35, 12 | 2.3 (62.37) | -5.8 (30.29)
  Week 21, On status, n=33, 11 | -0.1 (62.87) | -7.1 (36.34)
  Week 25, On status, n=33, 12 | -1.7 (41.50) | -0.7 (46.77)
  Week 37, On status, n=26, 12 | 8.0 (64.38) | -8.6 (34.96)
  Week 49, On status, n=20, 9 | 27.8 (99.17) | 1.8 (54.21)
  Week 52, On status, n=19, 9 | 7.5 (93.46) | 0.7 (54.13)
  Week 17, Off status, n=26, 13 | -1.4 (29.10) | -3.6 (14.44)
  Week 21, Off status, n=24, 12 | -4.4 (35.76) | -6.0 (9.09)
  Week 25, Off status, n=24, 13 | 1.4 (41.65) | -5.2 (38.30)
  Week 37, Off status, n=20, 13 | 6.1 (54.09) | 6.3 (50.27)
  Week 49, Off status, n=16, 11 | 1.9 (41.71) | 44.5 (96.82)
  Week 52, Off status, n=15, 11 | 7.1 (39.24) | 26.2 (50.57)

17. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 3 Total Score at the Indicated Visits in the Long Term Phase
Description: The Japanese UPDRS assessed the status of PD participants objectively. Part 3 evaluated motor examination on 27 items, response for each items were scored numerically from 0-4. The total score for the 27 items ranged from 0 to 108. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Percent change
  Week 17, n=41, 16 | -5.4 (20.98) | 6.2 (38.25)
  Week 21, n=39, 16 | -10.5 (25.83) | -6.0 (35.72)
  Week 25, n=40, 17 | -10.3 (31.99) | 2.6 (36.71)
  Week 37; n=33, 17 | -6.4 (30.91) | 50.2 (148.56)
  Week 49; n=26, 14 | -3.4 (46.73) | 43.2 (134.85)
  Week 52; n=25, 14 | -4.1 (44.35) | 16.2 (77.23)

18. Secondary Outcome: Percent Change From Baseline in the Japanese UPDRS Part 4 Total Score at the Indicated Visits in the Long-term Phase
Description: The Japanese UPDRS assesses the status of PD participants objectively. Part 4 evaluates complications on 11 items, response for 4 items were scored numerically from 0-4 and response for other 7 items were Yes/No questions and responses are numerically scored as 0 for "No" and 1 for "Yes". The total score for the 11 items ranged from 0 to 23. A higher score indicates more severe PD symptoms. Percent change from Baseline was calculated as Post baseline value minus Baseline value, divided by Baseline value and multiplied by 100. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Ropinirole CR - Maintenance Dose Group: Long Term Phase: Participants received ropinirole CR 16 mg administered orally OD for 4 weeks in the Screening Phase. After randomization participants entered Dose Increase Effect Verification Phase, where Ropinirole CR dose was maintained at 16 mg/day and the placebo was titrated to maintain blinding at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. This was followed by a down titration phase for one week and Long-term Phase for 39 weeks in which the participants received incremental doses (2 mg/day/week) of ropinirole CR from 18 mg/day to a maximum of 24 mg/day until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose. Participants completed the Long-term Phase underwent a down titration phase 2 for 1 to 2 weeks.
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Percent change
  Week 17, n=30, 15 | 13.1 (49.42) | 7.1 (43.29)
  Week 21, n=28, 14 | 11.3 (48.62) | 6.8 (41.68)
  Week 25, n=28, 15 | 16.4 (41.65) | 18.7 (101.42)
  Week 37, n=23, 15 | 11.3 (38.32) | 49.5 (139.78)
  Week 49, n=18, 13 | 27.5 (34.93) | 40.0 (123.78)
  Week 52, n=17, 13 | 23.7 (36.32) | 35.4 (104.67)

19. Secondary Outcome: Change From Baseline in the Actual Hours of Awake Time Spent "Off" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Change from Baseline in awake time spent "Off"(actual hours) is calculated as awake time spent "Off" (hours) at the indicated visit minus awake time spent "Off" (hours) at Baseline. Baseline is defined as the value at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 46 | 13
hours
  Week 2 | 0.14 (2.260) | 0.44 (1.605)
  Week 4 | 0.09 (2.308) | 0.04 (1.817)
  Week 6 | 0.01 (2.645) | 0.37 (2.068)
  Week 8 | -0.08 (2.552) | 0.77 (2.442)
  Week 12 | -0.27 (2.781) | 0.81 (1.953)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.65 to 1.04] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "Off" for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-1.34 to 1.45] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "Off" for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.95 to 1.24] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "Off" for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-2.44 to 0.75] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "Off" for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-2.73 to 0.58] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "Off" for Week 12

20. Secondary Outcome: Change From Baseline in the Percentage of Awake Time Spent "Off" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Percentage of awake time spent "off" is defined as sum of two days off time (hours) divided by sum of two days awake time (hours) and multiplied by 100. Change from Baseline was calculated by subtracting the Baseline value (percentage of awake time spent "off") from the post Baseline value (percentage of awake time spent "off"). Baseline is defined as the value at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: FAS1 Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of awake time spent off
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 46 | 13
percentage of awake time spent off
  Week 2 | 1.36 (13.025) | 2.39 (9.119)
  Week 4 | 0.62 (13.486) | 0.48 (10.116)
  Week 6 | -0.09 (15.677) | 2.70 (10.518)
  Week 8 | 0.19 (16.012) | 4.65 (12.040)
  Week 12 | -1.24 (16.814) | 4.74 (11.214)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-8.77 to 6.71] — Estimated value and CI are presented for the change from Baseline in the proportion of awake time spent "Off" for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-7.94 to 8.22] — Estimated value and CI are presented for the change from Baseline in the proportion of awake time spent "Off" for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -2.78, 95% CI 2-sided [-12.06 to 6.49] — Estimated value and CI are presented for the change from Baseline in the proportion of awake time spent "Off" for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -4.46, 95% CI 2-sided [-14.06 to 5.14] — Estimated value and CI are presented for the change from Baseline in the proportion of awake time spent "Off" for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = -5.98, 95% CI 2-sided [-15.92 to 3.96] — Estimated value and CI are presented for the change from Baseline in the proportion of awake time spent "Off" for Week 12

21. Secondary Outcome: Change From Baseline in Actual Hours of Awake Time Spent "On" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Change from Baseline in awake time spent "On"(actual hours) is calculated as awake time spent "On" (hours) at the indicated visit minus awake time spent "On" (hours) at Baseline. Baseline is defined as the value at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 53 | 18
hours
  Week 2, n=53, 17 | -0.39 (2.154) | -0.46 (1.635)
  Week 4, n=53, 18 | -0.12 (2.271) | -0.60 (2.180)
  Week 6, n=53, 18 | -0.01 (2.474) | -0.61 (1.676)
  Week 8, n=53, 18 | -0.11 (2.759) | -0.96 (1.554)
  Week 12, n=53, 18 | 0.07 (2.789) | -0.79 (1.815)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.07 to 1.21] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.75 to 1.70] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-0.65 to 1.86] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.52 to 2.22] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-0.55 to 2.26] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" for Week 12

22. Secondary Outcome: Change From Baseline in Actual Hours of Awake Time Spent "On"Without Troublesome Dyskinesias at the Indicated Visits Only in Participants Who Received L-dopa Adjunct
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Change from Baseline in awake time spent "On" without troublesome dyskinesias (actual hours) is calculated as [awake time spent "On" minus awake time spent "On" with troublesome dyskinesias] (hours) at visit minus [awake time spent "On" minus awake time spent "On" with troublesome dyskinesias] (hours) at Baseline. Baseline is defined as the value at Week 0. The analyses for Dose Increase Effect Verification Phase was performed using the LOCF data. In the LOCF data, the last available data was used for the imputation for missing data at a planned visit.
Time Frame: Baseline, Weeks, 2, 4, 6, 8 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 53 | 18
hours
  Week 2, n=53, 17 | -0.40 (2.276) | -0.59 (1.400)
  Week 4, n=53, 18 | -0.14 (2.359) | -0.71 (1.745)
  Week 6, n=53, 18 | -0.06 (2.566) | -0.63 (1.476)
  Week 8, n=53, 18 | -0.05 (2.896) | -1.01 (1.549)
  Week 12, n=53, 18 | 0.11 (2.968) | -0.74 (1.733)
Statistical Analysis 1: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.98 to 1.36] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" without troublesome dyskinesias for Week 2
Statistical Analysis 2: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.64 to 1.78] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" without troublesome dyskinesias for Week 4
Statistical Analysis 3: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.71 to 1.84] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" without troublesome dyskinesias for Week 6
Statistical Analysis 4: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [-0.47 to 2.39] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" without troublesome dyskinesias for Week 8
Statistical Analysis 5: Comparison: Ropinirole CR - High Dose Group vs Ropinirole CR - Maintenance Dose Group; Test type: Superiority or Other; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-0.63 to 2.33] — Estimated value and CI are presented for the change from Baseline in actual hours of awake time spent "On" without troublesome dyskinesias for Week 12

23. Secondary Outcome: Number of Participants With an Improvement (Responder) in the Clinical Global Impression (CGI) Global Improvement Scale at Week 12
Description: The CGI global improvement scale allows the investigator to rate the participant's total improvement since the beginning of treatment (Baseline). Scores on the scale range from 1 to 7 (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse). Participants with a CGI global improvement score of <=2 (representing much improved or very much improved) were considered to be moderate improvement (responder). The analyses performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Week 12
Population: FAS1 Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 52 | 19
Participants | 19 | 6

24. Secondary Outcome: Number of Participants Remaining in the Study
Time Frame: From the start of the study medication (Week 0) until Week 52
Population: Safety Population 2 (SP2) compraised of all participants who included in SP1 (receive at least one dose of medication in Dose Increase Effect Verification Phase) and shifted to Long-term Phase and received at least one dose of medication in Long-term Phase.
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Dose Group
Number analyzed (Participants) | 44 | 18
Participants | 25 | 14

25. Secondary Outcome: Number of Participants Achieving a 30% and 20% Reduction From Baseline in the UPDRS Total Part 3 Score at the Indicated Visits in Long Term Phase.
Description: The Japanese UPDRS assesses the status of Parkinson's Disease (PD) participants objectively. Part III assessed motor examination on 27 items. Participants received a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms. Number of participants achieving a 30% or greater and 20% or greater reduction from Baseline in UPDRS total part III score at Weeks 17, 21, 25, 37, 49 and 52,are presented using OC data. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline value. Baseline is defined as the value evaluated at Week 13. If the value evaluated at Week 13 was missing, then first observed value post Week 13 was used as Baseline. The OC (observed Case) dataset was defined as the dataset consisting of observed data without any missing data imputation.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49, 52
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Number analyzed (Participants) | 44 | 17
Participants
  Week 17, >=30% reduction from Baseline; n=41,16 | 5 | 2
  Week 21, >=30% reduction from Baseline; n=39,16 | 8 | 3
  Week 25, >=30% reduction from Baseline; n=40, 17 | 9 | 3
  Week 37, >=30% reduction from Baseline; n=33,17 | 8 | 3
  Week 49, >=30% reduction from Baseline; n=26, 14 | 9 | 1
  Week 52, >=30% reduction from Baseline; n=25, 14 | 6 | 2
  Week 17, >=20% reduction from Baseline; n=41,16 | 8 | 2
  Week 21, >=20% reduction from Baseline; n=39,16 | 15 | 3
  Week 25, >=20% reduction from Baseline; n=40, 17 | 16 | 3
  Week 37, >=20% reduction from Baseline; n=33,17 | 14 | 3
  Week 49, >=20% reduction from Baseline; n=26, 14 | 13 | 3
  Week 52, >=20% reduction from Baseline; n=25, 14 | 12 | 4

26. Secondary Outcome: Change From Baseline in the Actual Hours of Awake Time Spent "Off" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct in Long Term Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Change from Baseline was calculated by subtracting the Baseline value (actual hours of awake time spent "off") from the week 17, 21, 25, 37, 49 and 52 value (proportion of awake time spent "off"). Baseline is defined as the value at Week 13. If the value evaluated at week 13 was missing then first observed value post week 13 was used as a Baseline.The analyses for long term phase was performed using the OC data. In the OC data, no imputation was carried for any missing data
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: FAS2 Population who received L-dopa adjunct in Long term phase. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the FAS2 population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 38 | 15
hours
  Week 17, n=26, 13 | -0.63 (2.600) | -0.50 (1.829)
  Week 21, n=24, 12 | -0.40 (1.892) | -0.65 (1.428)
  Week 25, n=24, 13 | 0.04 (1.442) | -0.52 (1.325)
  Week 37, n=20, 13 | 0.01 (2.999) | -0.46 (2.252)
  Week 49, n=18, 11 | -0.24 (1.945) | 0.91 (3.117)
  Week 52, n=15, 11 | -0.62 (1.797) | 0.45 (2.255)

27. Secondary Outcome: Change From Baseline in the Percentage of Awake Time Spent "Off" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct in Long Term Phase
Description: "Off" state is defined as the state at which PD symptoms are not adequately controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Percentage of awake time spent "off" is defined as sum of two days off time (hours) divided by sum of two days awake time (hours) and multiplied by 100. Change from Baseline was calculated by subtracting the Baseline value (percentage of awake time spent "off") from week 17, 21, 25, 37, 49 and 52 value (percentage of awake time spent "off"). Baseline is defined as the value at Week 13, If the value evaluated at week 13 was missing then first observed value post week 13 was used as a Baseline. The analyses for Long term phase was performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of awake time spent off
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 38 | 15
percentage of awake time spent off
  Week 17, n=26, 13 | -4.16 (15.734) | -4.41 (16.606)
  Week 21, n=24, 12 | -2.59 (10.682) | -5.39 (13.102)
  Week 25, n=24, 13 | 0.49 (8.123) | -3.95 (10.677)
  Week 37, n=20, 13 | -0.99 (15.204) | -4.56 (20.134)
  Week 49, n=18, 11 | -1.33 (11.509) | 2.93 (19.464)
  Week 52, n=15, 11 | -3.62 (9.925) | 1.24 (13.957)

28. Secondary Outcome: Change From Baseline in Actual Hours of Awake Time Spent "On" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct in Long Term Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Participants were asked to record the duration of their "off " periods and asleep in diary cards every day. Change from Baseline in awake time spent "On"(actual hours) is calculated as awake time spent "On" (hours) at the week 17, 21, 25, 37, 49 and 52 value minus awake time spent "On" (hours) at Baseline. Baseline is defined as the value at Week 13. If the value evaluated at week 13 was missing then first observed value post week 13 was used as a Baseline. The analyses for Long term phase was performed using the OC data. The OC (observed Case) dataset was defined as the dataset consisting of observed data without any missing data imputation.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 38 | 15
hours
  Week 17, n=36, 15 | 0.56 (2.472) | 0.57 (2.376)
  Week 21, n=34, 14 | 0.43 (1.585) | 0.73 (2.006)
  Week 25, n=34, 15 | -0.04 (1.434) | 0.23 (1.896)
  Week 37, n=29, 15 | 0.26 (2.188) | 0.37 (3.266)
  Week 49, n=26, 12 | -0.19 (1.764) | -0.56 (3.163)
  Week 52, n=23, 12 | 0.36 (1.539) | -0.56 (2.358)

29. Secondary Outcome: Change From Baseline in Actual Hours of Awake Time Spent "On" Without Troublesome Dyskinesias at the Indicated Visits Only in Participants Who Received L-dopa Adjunct in Long Term Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Participants were asked to record the duration of their "on " periods and asleep in diary cards every day. Change from Baseline in awake time spent "On" without troublesome dyskinesias (actual hours) is calculated as [awake time spent "On" minus awake time spent "On" with troublesome dyskinesias] (hours) at visit minus [awake time spent "On" minus awake time spent "On" with troublesome dyskinesias] (hours) at Baseline. Baseline is defined as the value at Week 13. If the value evaluated at week 13 was missing then first observed value post week 13 was used as a Baseline. The analyses for Long term phase was performed using the OC data. In the OC data, no imputation was carried for any missing data
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 38 | 15
hours
  Week 17, n=36, 15 | 0.24 (2.245) | 0.60 (2.347)
  Week 21, n=34, 14 | 0.21 (1.850) | 1.23 (2.403)
  Week 25, n=34, 15 | -0.15 (1.341) | 0.25 (2.615)
  Week 37, n=29, 15 | -0.09 (2.247) | 1.02 (3.447)
  Week 49, n=26, 12 | -0.50 (1.877) | 0.04 (2.720)
  Week 52, n=23, 12 | 0.08 (1.378) | -0.21 (2.886)

30. Secondary Outcome: Change From Baseline in Percentage of Awake Time Spent "On" at the Indicated Visits Only in Participants Who Received L-dopa Adjunct in Long Term Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Participants were asked to record the duration of their "on " periods and asleep in diary cards every day. Percentage of awake time spent "on" is defined as sum of two days on time (hours) divided by sum of two days awake time (hours) and multiplified by 100. Change from Baseline was calculated by subtracting the Baseline value (percentage of awake time spent "on") from week 17, 21, 25, 37, 49 and 52 value (percentage of awake time spent "on"). Baseline is defined as the value at Week 13. If the value evaluated at week 13 was missing the first observed value post week 13 was used as a Baseline.The analyses for Long term phase was performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of awake time spent on
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 38 | 15
percentage of awake time spent on
  Week 17, n=36, 15 | 2.81 (13.529) | 3.82 (15.452)
  Week 21, n=34, 14 | 1.20 (9.841) | 4.62 (12.211)
  Week 25, n=34, 15 | -1.02 (7.813) | 3.42 (9.982)
  Week 37, n=29, 15 | 0.13 (12.766) | 3.27 (19.048)
  Week 49, n=26, 12 | -0.23 (10.389) | -2.68 (18.578)
  Week 52, n=23, 12 | 1.80 (8.706) | -1.14 (13.313)

31. Secondary Outcome: Change From Baseline in Percentage of Awake Time Spent "On" Without Troublesome Dyskinesias at the Indicated Visits Only in Participants Who Received L-dopa Adjunct in Long Term Phase
Description: "On" state is defined as the state at which PD symptoms are well controlled by the drug. Par. were asked to record the duration of their "on " periods and asleep in diary cards every day. Percentage of awake time spent "On" without troublesome dyskinesias is defined as sum of two days on time without troublesome dyskinesias ["On" time minus "On" time with troublesome dyskinesias] (hours) divided by sum of two days awake time (hours) and multiplified by 100. Change from Baseline was calculated by subtracting the Baseline value (percentage of awake time spent "On" without troublesome dyskinesias) from week 17, 21, 25, 37, 49 and 52 value (percentage of awake time spent "On" without troublesome dyskinesias). Baseline is defined as the value at Week 13. If the value evaluated at week 13 was missing the first observed value post week 13 was used as a Baseline.The analyses for Long term phase was performed using the OC data. In the OC data, no imputation was carried for any missing data.
Time Frame: Baseline (Week 13), Weeks 17, 21, 25, 37, 49 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percentage of awake time spent on
Arm/Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Dose Group: Long Term Phase
Number analyzed (Participants) | 38 | 15
percentage of awake time spent on
  Week 17, n=36, 15 | 0.70 (11.655) | 4.04 (15.472)
  Week 21, n=34, 14 | -0.16 (11.730) | 7.31 (13.780)
  Week 25, n=34, 15 | -1.70 (7.765) | 3.10 (15.036)
  Week 37, n=29, 15 | -1.71 (13.698) | 6.93 (19.472)
  Week 49, n=26, 12 | -2.00 (11.835) | 0.45 (15.958)
  Week 52, n=23, 12 | -0.05 (7.521) | 0.53 (14.966)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected from the start of study treatment (Week 0) until Week 52.
Description: SAEs and non-SAEs were collected in participants of the SP1 Population, comprised of all participants who had received at least one dose of medication in the Dose Increase Effect Verification Phase.
Groups:
- Ropinirole CR - Maintenance Group; Ropinirole CR - Maintenance Group: Long Term Phase: Participants received ropinirole CR 16 mg administered orally OD for 4 weeks in the Screening Phase. After randomization participants entered Dose Increase Effect Verification Phase, where Ropinirole CR dose was maintained at 16 mg/day and the placebo was titrated to maintain blinding at intervals of 1 week or longer for 8 weeks, until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose for 4 weeks. This was followed by a down titration phase for one week and Long-term Phase for 39 weeks in which the participants received incremental doses (2 mg/day/week) of ropinirole CR from 18 mg/day to a maximum of 24 mg/day until participants reached a dose level above which further symptomatic improvement was not expected; the participants were maintained on that dose. Participants completed the Long-term Phase underwent a down titration phase 2 for 1 to 2 weeks.
Arm/Group | Ropinirole CR - High Dose Group | Ropinirole CR - Maintenance Group | Ropinirole CR - High Dose Group: Long Term Phase | Ropinirole CR - Maintenance Group: Long Term Phase
Serious Adverse Events (participants affected / at risk) | 2/61 | 4/20 | 0/44 | 1/18
Other Adverse Events (participants affected / at risk) | 13/61 | 11/20 | 14/44 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole CR - High Dose Group (N=61) | Ropinirole CR - Maintenance Group (N=20) | Ropinirole CR - High Dose Group: Long Term Phase (N=44) | Ropinirole CR - Maintenance Group: Long Term Phase (N=18)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ropinirole CR - High Dose Group (N=61) | Ropinirole CR - Maintenance Group (N=20) | Ropinirole CR - High Dose Group: Long Term Phase (N=44) | Ropinirole CR - Maintenance Group: Long Term Phase (N=18)
Dyskinesia (Nervous system disorders) | 3 | 2 | 2 | 1
Somnolence (Nervous system disorders) | 4 | 1 | 0 | 0
Sudden onset of sleep (Nervous system disorders) | 2 | 2 | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 4 | 5 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 2
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Sleep attacks (Psychiatric disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.